CLINICAL TRIAL: NCT03572400
Title: Neoadjuvant CCRT With Gemcitabine/Durvalumab (MEDI4736) Followed by Adjuvant Gemcitabine/Durvalumab(MEDI4736) in Resectable or Borderline Resectable Pancreatic Cancer
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Do-Youn Oh (Other)
Collaborators: AstraZeneca (Industry)
Responsible Party: Sponsor-Investigator, Do-Youn Oh, Professor, Seoul National University Hospital
Organization: Seoul National University Hospital (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ESR-16-12315
Record Dates: First submitted 2018-06-18; First posted 2018-06-28 (Actual); Last update posted 2024-04-19 (Actual); Status verified 2024-04

CONDITIONS: Pancreatic Cancer
Keywords: pancreatic cancer; pancreas cancer
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Gemcitabine; durvalumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Gemcitbine/Durvalumab (Experimental): Neoadjuvant CCRT with Gemcitbine/Durvalumab
  +Adjuvant Gemcitabine/Durvalumab Total 6 cycles, after that, Durvalumab q4wks up to total 1 year
  Interventions: Drug: Gemcitabine; Drug: Durvalumab

INTERVENTIONS:
Drug: Gemcitabine — Neoadjuvant: Weekly Gemcitabine 200 mg/m2 iv Adjuvant: Gemcitabine 1000mg/m2, D1, 8, 15 Q 4 weeks total 6cycles
Drug: Durvalumab — Neoadjuvant: Durvalumab 1.5g iv Q 4weeks Adjuvant: Durvalumab 1.5g iv Q 4weeks for 1 year

SUMMARY:
<Research Hypothesis> The dynamics of immune cells by CCRT/Durvalumab will be uncovered. The combination of Durvalumab with concurrent chemoradiotherapy (CCRT/gemcitabine)) as neoaduvant treatment in resectable or borderline resectable pancreatic cancer is feasible and efficacious.

The combination of Durvalumab with cytotoxic chemotherapy (gemcitabine) as an adjuvant treatment is feasible and efficacious.

<Objectives> To assess the effect of Neoadjuvant CCRT with Gemcitabine/Durvalumab followed by adjuvant Gemcitabine/Durvalumab in resectable or borderline resectable pancreatic cancer

Primary endpoint:

2 year-DFSR (disease-free survival rate) Secondary endpoints

* Efficacy: 2 year-OSR (overall survival rate), disease-free survival, overall survival, overall response rate (RECIST 1.1, ir response) after neoadjuvant CCRT, disease control rateEORTC QLQ-C30, the number of immune cells (TIL, macrophage, etc) in resected pancreatic tissue
* Safety: toxicity (CTCAE V), irAE,

Exploratory Objective(s):

* To evaluate baseline measures and changes of immune systems and regulations by neoadjuvant CCRT with gemcitabine/Durvalumab in peripheral blood and tumor tissues
* To collect and store DNA from blood (according to ethical procedures) for future exploratory research into genes/genetic variation that may influence response (ie, distribution, safety, tolerability and efficacy) to study treatments and or susceptibility to disease (optional).

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent and any locally-required authorization (eg, HIPAA in the USA, EU Data Privacy Directive in the EU) obtained from the subject prior to performing any protocol-related procedures, including screening evaluations
2. Age>=19 years at time of study entry
3. Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1
4. Life expectancy of >= 3months
5. Histologically proven pancreatic ductal adenocarcinoma
6. Resectable or borderline resectable based on AJCC Cancer staging system (8th ed)
7. Chemotherapy -naïve for their pancreatic cancer
8. Body weight >30kg (for durvalumab monotherapy or durvalumab + novel)
9. Adequate normal organ and marrow function as defined below: (NOTE TO AUTHOR: These are minimum criteria for studies in subjects with solid tumors and may need to be altered based on individual study requirements; please adjust as necessary) -Haemoglobin ≥ 9.0 g/dL

   * Absolute neutrophil count (ANC) 1.5 (or 1.0) x (> 1500 per mm3)
   * Platelet count ≥ 100 (or 75) x 109/L (>75,000 per mm3)
   * Serum bilirubin ≤ 1.5 x institutional upper limit of normal (ULN). This will not apply to subjects with confirmed Gilbert's syndrome (persistent or recurrent hyperbilirubinemia that is predominantly unconjugated in the absence of hemolysis or hepatic pathology), who will be allowed only in consultation with their physician.
   * AST (SGOT)/ALT (SGPT) ≤ 2.5 x institutional upper limit of normal unless liver metastases are present, in which case it must be ≤ 5x ULN
   * Serum creatinine CL>40 mL/min by the Cockcroft-Gault formula (Cockcroft and Gault 1976) or by 24-hour urine collection for determination of creatinine clearance:
10. Evidence of post-menopausal status or negative urinary or serum pregnancy test for female pre-menopausal subjects. Women will be considered post-menopausal if they have been amenorrheic for 12 months without an alternative medical cause. The following age-specific requirements apply:
11. Subject is willing and able to comply with the protocol for the duration of the study including undergoing treatment and scheduled visits and examinations including follow up.

Exclusion Criteria:

25. Participation in another clinical study with an investigational product during the last 3 weeks 26. Concurrent enrolment in another clinical study, unless it is an observational (non-interventional) clinical study or during the follow-up period of an interventional study 27. Any previous treatment with a PD1 or PD-L1 inhibitor, including durvalumab 28. Receipt of the last dose of anti-cancer therapy (chemotherapy, immunotherapy, endocrine therapy, targeted therapy, biologic therapy, tumor embolization, monoclonal antibodies, other investigational agent) 28 days prior to the first dose of study drug 29. Mean QT interval corrected for heart rate (QTc) ≥470 ms calculated from 3 electrocardiograms (ECGs) using Fridericia's Correction (this can be removed if testing durvalumab alone and retain this exclusion if combining durvalumab with novel agents) 30. Current or prior use of immunosuppressive medication within 14days (use 28 days if combining durvalumab with a novel agent) before the first dose of durvalumab, with the exceptions of intranasal and inhaled corticosteroids or systemic corticosteroids at physiological doses, which are not to exceed 10 mg/day of prednisone, or an equivalent corticosteroid. The following are exceptions to this criterion:

- Intranasal, inhaled, topical steroids, or local steroid injections (eg, intra articular injection)

* Systemic corticosteroids at physiologic doses not to exceed <<10 mg/day>> of prednisone or its equivalent
* Steroids as premedication for hypersensitivity reactions (eg, CT scan premedication) 31. Any unresolved toxicity NCI CTCAE Grade ≥2 from previous anticancer therapy with the exception of alopecia, vitiligo, and the laboratory values defined in the inclusion criteria
* Subjects with Grade ≥2 neuropathy will be evaluated on a case-by-case basis after consultation with the Study Physician.
* Subjects with irreversible toxicity not reasonably expected to be exacerbated by treatment with durvalumab may be included only after consultation with the Study Physician.

  32. Any concurrent chemotherapy, IP, biologic, or hormonal therapy for cancer treatment. Concurrent use of hormonal therapy for non-cancer-related conditions (eg, hormone replacement therapy) is acceptable. <<amend as required based on any combination studies with other anti-cancer agents>> 33. <<if applicable to the study>>Radiotherapy treatment to more than 30% of the bone marrow or with a wide field of radiation within 4 weeks of the first dose of study drug 34. Major surgical procedure (as defined by the Investigator) within 28 days prior to the first dose of IP. Note: Local surgery of isolated lesions for palliative intent is acceptable.

  35. History of allogenic organ transplantation. 36. Active or prior documented autoimmune or inflammatory disorders (including inflammatory bowel disease [eg, colitis or Crohn's disease], diverticulitis [with the exception of diverticulosis], systemic lupus erythematosus, Sarcoidosis syndrome, or Wegener syndrome [granulomatosis with polyangiitis, Graves' disease, rheumatoid arthritis, hypophysitis, uveitis, etc]). The following are exceptions to this criterion:
* Subjects with vitiligo or alopecia
* Subjects with hypothyroidism (eg, following Hashimoto syndrome) stable on hormone replacement
* Any chronic skin condition that does not require systemic therapy
* Subjects without active disease in the last 5 years may be included but only after consultation with the study physician
* Subjects with celiac disease controlled by diet alone 37. Uncontrolled intercurrent illness, including but not limited to, ongoing or active infection, symptomatic congestive heart failure, uncontrolled hypertension, unstable angina pectoris, cardiac arrhythmia, interstitial lung disease, serious chronic gastrointestinal conditions associated with diarrhea, or psychiatric illness/social situations that would limit compliance with study requirement, substantially increase risk of incurring AEs or compromise the ability of the patient to give written informed consent 38. History of another primary malignancy except for
* Malignancy treated with curative intent and with no known active disease ≥5 years before the first dose of IP and of low potential risk for recurrence
* Adequately treated non-melanoma skin cancer or lentigo maligna without evidence of disease
* Adequately treated carcinoma in situ without evidence of disease 39. History of leptomeningeal carcinomatosis 40. Brain metastases or spinal cord compression. 41. Mean QT interval corrected for heart rate using Fridericia's formula (QTcF) ≥470 ms calculated from 3 ECGs (within 15 minutes at 5 minutes apart) <<for durvalumab monotherapy and durvalumab + tremelimumab combination studies this criterion can be removed. For durvalumab ± tremelimumab in combination with an agent with pro-arrhythmic potential or where effect of the combination on QT is not known if this criterion should be retained. Patient safety and the cardiac SKG should be consulted as needed>>.

  42. History of active primary immunodeficiency 43. Active infection including tuberculosis (clinical evaluation that includes clinical history, physical examination and radiographic findings, and TB testing in line with local practice), hepatitis B (known positive HBV surface antigen (HBsAg) result), hepatitis C, or human immunodeficiency virus (positive HIV 1/2 antibodies). Subjects with a past or resolved HBV infection (defined as the presence of hepatitis B core antibody [anti-HBc] and absence of HBsAg) are eligible. Subjects positive for hepatitis C (HCV) antibody are eligible only if polymerase chain reaction is negative for HCV RNA.

  44. Current or prior use of immunosuppressive medication within 14 days before the first dose of durvalumab or tremelimumab. The following are exceptions to this criterion:
* Intranasal, inhaled, topical steroids, or local steroid injections (eg, intra articular injection)
* Systemic corticosteroids at physiologic doses not to exceed <<10 mg/day>> of prednisone or its equivalent
* Steroids as premedication for hypersensitivity reactions (eg, CT scan premedication) 45. Receipt of live attenuated vaccine within 30 days prior to the first dose of IP. Note: Subjects, if enrolled, should not receive live vaccine whilst receiving IP and up to 30 days after the last dose of IP.

  46. Female subjects who are pregnant or breastfeeding or male or female subjects of reproductive potential who are not willing to employ effective birth control from screening to 90 days after the last dose of durvalumab monotherapy.

  47. Known allergy or hypersensitivity to any of the study drugs or any of the study drug excipients.

  48. Prior randomisation or treatment in a previous durvalumab and/or tremelimumab clinical study regardless of treatment arm assignment.

  49. Past medical history of ILD, drug-induced ILD, radiation pneumonitis which required steroid treatment, or any evidence of clinically active interstitial lung disease.

  50. Judgment by the investigator that the patient is unsuitable to participate in the study and the patient is unlikely to comply with study procedures, restrictions and requirements.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 71 (Estimated)
Dates: Start 2018-11-29 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Disease-free survival rate | 8 weeks
  The percentage of time from enroll until disease progression or death

SECONDARY OUTCOMES:
Overall survival | 12weeks
  Time from enroll until death from any cause
Disease-free survival | 8 weeks
  Time from enroll until disease progression or death
Overall response rate | 8 weeks
  RECIST 1.1, ir response
Safety and tolerability as measured by number and grade of toxicity events | 2 weeks
  CTCAE v4.03
Disease control rate | 8 weeks
  The percentage of patients who have achieved complete response, partial response and stable disease

CONTACTS AND LOCATIONS:
Overall Officials: Do-Youn Oh, MD, PhD, Principal Investigator — Seoul National University Hospital
Locations (1):
- Seoul National University Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No